CLINICAL TRIAL: NCT07027982
Title: An Open-label, Randomized, Single-dose, Crossover Study to Evaluate the Pharmacokinetics and Safety of Diluted vs. Undiluted Intravenous DA-5217 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of Diluted vs. Undiluted Intravenous DA-5217 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: DA5217_UGIB_I
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Healthy Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental)
  Interventions: Drug: Diluted Intravenous DA-5217; Drug: Undiluted Intravenous DA-5217
- Sequence 2 (Experimental)
  Interventions: Drug: Diluted Intravenous DA-5217; Drug: Undiluted Intravenous DA-5217

INTERVENTIONS:
Drug: Diluted Intravenous DA-5217 — once a day
Drug: Undiluted Intravenous DA-5217 — once a day

SUMMARY:
This study will evaluate the pharmacokinetics and safety of Diluted and Undiluted Intravenous DA-5217 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female, 19 years to 45 years
* Weighing 50 kg or more, with a body mass index (BMI) of 18.5 kg/m2 to 29.9kg/m2
* The subjects signed and dated informed consent form after hearing a detailed explanation of the study, fully understanding and determined voluntarily to participate and complied with the precautions.

Exclusion Criteria:

* The subjects with existing or previous conditions that may influence the pharmacokinetics of drugs
* The subjects hypersensitive to any of the Investigational Product components or other drug components
* The subjects with clinically significant active chronic conditions
* The subjects with a positive urine drug test result or a history of drug abuse or dependence.
* The subjects who are pregnant or lactating

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-07-16 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
AUClast | 0~24hours
  Area under the plasma concentration-time curve from time zero to time the last quantifiable time

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea